CLINICAL TRIAL: NCT01988233
Title: BAILA: Being Active, Increasing Latinos Healthy Aging
Acronym: BAILA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, David Xavier Marquez, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012-0851; 1R01NR013151 (NIH)
Record Dates: First submitted 2013-11-05; First posted 2013-11-20 (Estimated); Results first posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Mobility Limitation
Keywords: Physical activity; Dance; Latinos; Aging; Older adults; Health disparities
MeSH Terms: conditions — Mobility Limitation; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BAILAMOS© Dance Program (Experimental): BAILAMOS© Dance Program + Maintenance Program: includes a 4-month twice-weekly adoption phase and a 4-month twice-weekly maintenance phase. Each month during adoption a new dance style is introduced by a professional dance instructor. During the 4-month maintenance phase an indigenous dance leader, trained by the professional dance instructor, will lead dance with participants twice per week
  Interventions: Behavioral: BAILAMOS© Dance Program
- Health Education Control Group (Experimental): Health Education Control Group: Sedentary older Latinos randomly assigned to the health education control group will participate in classes developed for older adults and offered by the University of Illinois Extension. All classes are conducted in Spanish by extension staff using Spanish-language materials. Classes will meet one day per week for two hours, to provide equitable social contact as the treatment group.
  Interventions: Behavioral: Health Education Control Group

INTERVENTIONS:
Behavioral: BAILAMOS© Dance Program
  Arms: BAILAMOS© Dance Program
Behavioral: Health Education Control Group
  Arms: Health Education Control Group

SUMMARY:
Investigators propose a randomized controlled trial (RCT) to test the efficacy of the revised 4-month BAILAMOS© program for improving lifestyle PA and health outcomes (physical and cognitive function, self-reported functional limitations, disability) in sedentary older Latinos at risk for disability relative to an attention control group.

DETAILED DESCRIPTION:
Older Latinos comprised 7% of the older adult population in 2002, but are expected to constitute 20% by 2050. Physical activity (PA) can influence potential declines in the health outcomes of physical and cognitive function that lead to functional limitations (self-reported restrictions in performance) and disability (functional limitations placed in a social context). Unfortunately, Latinos aged 65-74 are 46% less likely to engage in leisure time PA than older non-Latino whites and little is known about PA maintenance among ethnic minorities compared to non-Latino whites. In part as a result of low levels of PA, the physical and cognitive function of older Latinos is poor relative to older non-Latino whites.

Participation in PA has substantial potential to help older Latinos maintain both physical and cognitive function as they age. Walking and dancing are the two most commonly reported forms of PA among older Latinos. However, urban older Latinos cite unsafe neighborhoods and extreme weather conditions as significant barriers to walking. Dance is a widely popular form of PA among Latinos of all ages, and holds considerable promise as a culturally appropriate form of PA that challenges individuals both physically and cognitively. To date, PA programs designed for older Latinos are lacking. BAILAMOS© is an innovative dance program that has been developed by Dr. Marquez (PI) based on focus group input from older community-dwelling Latinos and in collaboration with an accomplished Latin dance instructor.

Investigators propose a randomized controlled trial (RCT) to test the efficacy of the revised 4-month BAILAMOS© program for improving lifestyle PA and health outcomes (physical and cognitive function, self-reported functional limitations, disability) in sedentary older Latinos at risk for disability relative to an attention control group. Investigators will also test whether lifestyle PA and health outcomes can be maintained over an additional 4-months through BAILAMOS© maintenance activities, which include using indigenous dance leaders. This study will use an RCT (N=166 Treatment, 166 Control) with a health education control group that will allow investigators to examine the adoption of PA and its impact on health outcomes (first 4 months), and the short-term maintenance of PA and its impact on health outcomes (8 months) among older Latinos.

ELIGIBILITY:
Inclusion Criteria:

* age > 55 years old
* self-identification as Latino/Hispanic
* ability to speak Spanish
* participation in <3 day/week of aerobic exercise
* at risk for disability
* adequate cognitive status as assessed by the Mini Mental State Examination
* danced < 2 times/month over the past 12 months
* willingness to be randomly assigned to treatment or control group
* no plans to leave the country for more than two consecutive weeks over the next year

Exclusion Criteria:

* uncontrolled cardiovascular disease
* uncontrolled diabetes mellitus
* pacemaker in situ
* severe chronic obstructive pulmonary disease (COPD)
* recent healing or unhealed fracture(s)
* use of an assistance device to walk (cane, walker, or wheelchair)

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2013-03; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David X Marquez, PhD, Principal Investigator — University of Illinois at Chicago
Locations (12):
- United States (12):
  - West Suburban Senior Services, Inc, Bellwood, Illinois
  - Catholic Charities of the Archdioceses of Chicago St Mary of Celle Strengthening Center, Berwyn, Illinois
  - Pilsen Senior Center, Chicago, Illinois
  - Holy Cross/Immaculate Heart of Mary Parish, Chicago, Illinois
  - Villa Guadalupe Senior Services, Inc., Chicago, Illinois
  - Northwest (Copernicus) Regional Senior Center, Chicago, Illinois
  - Dance Academy of Salsa, Chicago, Illinois
  - West Town Senior Center, Chicago, Illinois
  - St. Agnes of Bohemia Parish, Chicago, Illinois
  - Southwest Senior Center, Chicago, Illinois
  - Kelvyn Park Senior Center, Chicago, Illinois
  - Our Lady of Mount Carmel, Melrose Park, Illinois

REFERENCES:
- [Derived] Lopez O, Kaushal N, Jaldin MA, Marquez DX. Latin Dance Effects on Cardiorespiratory Fitness and Physical Function in Middle-Aged and Older Latino Adults. J Aging Phys Act. 2023 Nov 21;32(2):163-171. doi: 10.1123/japa.2022-0415. Print 2024 Apr 1. PMID 37989134
- [Derived] Aguinaga S, Kaushal N, Balbim GM, Wilson RS, Wilbur JE, Hughes S, Buchner DM, Berbaum M, McAuley E, Vasquez PM, Marques IG, Wang T, Marquez DX. Latin Dance and Working Memory: The Mediating Effects of Physical Activity Among Middle-Aged and Older Latinos. Front Aging Neurosci. 2022 Apr 15;14:755154. doi: 10.3389/fnagi.2022.755154. eCollection 2022. PMID 35493932
- [Derived] Marquez DX, Wilbur J, Hughes S, Wilson R, Buchner DM, Berbaum ML, McAuley E, Aguinaga S, Balbim GM, Vasquez PM, Marques IG, Wang T, Kaushal N. BAILA: A Randomized Controlled Trial of Latin Dancing to Increase Physical Activity in Spanish-Speaking Older Latinos. Ann Behav Med. 2022 Nov 18;56(12):1231-1243. doi: 10.1093/abm/kaac009. PMID 35445687

RESULTS

PARTICIPANT FLOW:
Groups:
- BAILAMOS© Dance Program: BAILAMOS© Dance Program + Maintenance Program: includes a 4-month twice-weekly adoption phase and a 4-month twice-weekly maintenance phase. Each month during adoption a new dance style is introduced by a professional dance instructor. During the 4-month maintenance phase an indigenous dance leader, trained by the professional dance instructor, will lead dance with participants twice per week
  BAILAMOS© Dance Program
- Health Education Control Group: Health Education Control Group: Sedentary older Latinos randomly assigned to the health education control group will participate in classes developed for older adults and offered by the University of Illinois Extension. All classes are conducted in Spanish by extension staff using Spanish-language materials. Classes will meet one day per week for two hours, to provide equitable social contact as the treatment group.
  Health Education Control Group
Period: Overall Study
Arm/Group | BAILAMOS© Dance Program | Health Education Control Group
Started | 167 | 166
Completed | 103 | 115
Not Completed | 64 | 51
Not completed — Lost to Follow-up | 64 | 51

BASELINE CHARACTERISTICS:
Population: 333 participants were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | BAILAMOS© Dance Program | Health Education Control Group | Total
Number analyzed (Participants) | 167 | 166 | 333
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.14 (6.39) | 65.67 (7.68) | 64.91 (7.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 141 | 281
  Male | 27 | 25 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 167 | 166 | 333
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 167 | 166 | 333
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.47 (4.54) | 30.84 (5.05) | 31.15 (4.79)

OUTCOME MEASURES:

1. Primary Outcome: Minutes Per Week of Moderate to Vigorous Physical Activity
Description: CHAMPS PA Questionnaire assesses weekly frequency and duration of a variety of lifestyle physical activities that are meaningful and appropriate for older adults.
Time Frame: Change from baseline to post-intervention 4 months
Population: Those randomized to intervention or control group.
Measure: Mean (Standard Deviation); unit: Change in minutes/week
Arm/Group | BAILAMOS© Dance Program | Health Education Control Group
Number analyzed (Participants) | 167 | 166
Change in minutes/week | 156.84 (12.57) | 86.84 (43.9)

2. Secondary Outcome: Physical Function Performance as Assessed by Time of 400 Meter Walk
Description: 400 Meter walk
Time Frame: Change from baseline to post-intervention 4 months
Population: Participants randomized to each group with data at baseline.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | BAILAMOS© Dance Program | Health Education Control Group
Number analyzed (Participants) | 151 | 149
Seconds | -0.31 (8.51) | 2.48 (13.76)

3. Secondary Outcome: Cognitive Function
Description: Working Memory: The score is the number of correctly retrieved strings in each part of the Digit Span Test plus the number of correctly reordered strings from the Digit Ordering. Higher scores indicated better outcomes. Higher change indicate better outcomes.
Time Frame: Change from baseline to post-intervention 4 months
Population: Data from participants randomized who had baseline data.
Measure: Mean (Standard Deviation); unit: Items recalled correctly
Arm/Group | BAILAMOS© Dance Program | Health Education Control Group
Number analyzed (Participants) | 167 | 166
Items recalled correctly | .25 (1.43) | .03 (1.44)

4. Secondary Outcome: Self-Reported Functional Limitations
Description: Function Subscale of Late Life Function & Disability Instrument. Higher scores reflect more limitation in performing tasks. Range on questionnaire is 15-75. Change is reported here.
Time Frame: Change from baseline to post-intervention 4 months
Population: Data from participants randomized at baseline who have baseline data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BAILAMOS© Dance Program | Health Education Control Group
Number analyzed (Participants) | 165 | 166
score on a scale | -0.51 (9.12) | 0.23 (8.12)

ADVERSE EVENTS:
Time Frame: The specific period of time over which adverse event data were collected was 1 year for each participant.
Description: All adverse events or unanticipated problems were to be reported in writing to the University Institutional Review Board within 5 days of the discovery. Serious or unexpected adverse events were to be verbally reported within 24 to 48 h.
Arm/Group | BAILAMOS© Dance Program | Health Education Control Group
All-Cause Mortality (participants affected / at risk) | 0/167 | 0/166
Serious Adverse Events (participants affected / at risk) | 0/167 | 0/166
Other Adverse Events (participants affected / at risk) | 0/167 | 0/166

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-06): https://cdn.clinicaltrials.gov/large-docs/33/NCT01988233/Prot_SAP_000.pdf